CLINICAL TRIAL: NCT03913286
Title: Neuromotor Prosthetic to Treat Stroke-Related Paresis
Acronym: Cortimo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 17D.459
Record Dates: First submitted 2019-03-07; First posted 2019-04-12 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Stroke, Complication; Stroke; Stroke Sequelae; Hemiparesis; Arm Paralysis
Keywords: neuroprosthetic; neuroprosthesis; brain-computer; brain-machine; microelectrode; Utah array; orthosis; brain computer interface; assistive device; Neurorehabilitation; neurotechnology
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention (Experimental): The participant will be implanted with the Blackrock Microsystems MultiPort system.
  Interventions: Device: Cortimo

INTERVENTIONS:
Device: Cortimo — The Cortimo comprises an implanted brain activity sensor and a wearable powered arm orthosis.
  Other Names: MyoPro powered orthotic brace; Blackrock Microsystems MultiPort

SUMMARY:
The purpose of the research is to develop a new medical device prototype to restore functional movement of an arm made weak due to a chronic stroke

DETAILED DESCRIPTION:
Microelectrode arrays implanted into the brain will decode signals to drive motors on the powered brace worn on the arm so that the patient can "power steer" his or her own arm. The ultimate goal is to create a fully implantable medical device that will restore movement in all parts of the body affected by a stroke. Independent movement will have functional benefits (e.g., being able to lift a fork to eat) and health benefits (e.g., decreasing the frequency of skin infections and preventing the formation of painful joint contractures).

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years or older.
* Clinical diagnosis of stroke (hemorrhagic or ischemic, cortical or subcortical), confirmed by brain computer tomography or magnetic resonance imaging, that occurred six or more months prior to enrollment
* Must have arm weakness due to stroke.
* Participant is willing to comply with all follow-up evaluations at the specified times.
* Participant is able to provide informed consent prior to enrollment in the study.
* The participant is fluent in English.
* > 24 on the Mini Mental Status Examination
* Medically stable.
* Passive flexion of shoulder in weakened upper extremity with range of > 30 degrees or more
* Passive abduction of shoulder in weakened upper extremity with range of > 20 degrees or more
* Participant must have a caregiver willing to participate in the study who will help provide care for the surgical site.
* Must be willing to live at hospital or at nearby hotel for 90-day duration when implantable components were present.
* Plateaued post-stroke recovery with complete or incomplete hemiplegia due to stroke in one upper limb, as measured on two serial occasions (at least one month apart) without improvement, by the following standardized functional assessments of the weaker upper extremity, at their worst:

  * Manual Muscle Testing scores of 0/5 (no movement) or 1/5 (palpable contraction in muscle, without movement) in the biceps (elbow flexion), triceps (elbow extension), wrist flexors, wrist extensors or intrinsic hand muscles
  * Mild to plegia according to Medical Research Council Scale for Muscle Strength
  * Fugl-Meyer Motor Impairment Score of 38 or lower
  * Action Research Arm Test (ARAT) score of 35 or lower
  * Motricity Index score of 55 or lower
* No joint contracture or severe spasticity in affected upper limb precluding the operation of the MyoPro orthotic device.
* Sufficient sitting balance to participate with robotic brace activities.
* No condition (e.g., severe arthritis, central pain) that would interfere with administration of motor function tests, ability to understand verbal commands and cooperate with test procedures.

Exclusion Criteria:

* No medical condition requiring active anti-coagulation with a medication such as heparin, warfarin or rivaroxaban (note that anti-platelet agents such as aspirin or clopidogrel are acceptable)
* No active wound healing or skin breakdown issues.
* No history of poorly controlled autonomic dysreflexia.
* Visual impairment such that extended viewing of a computer monitor would be challenging even with ordinary corrective lenses
* Chronic oral or intravenous steroids or immunosuppressive therapy
* A score of 23 or lower on Folstein's Mini-Mental Status Examination
* Orthopedic conditions of either arm that would affect performance on study
* Untreated psychiatric disturbances that would affect motivation and trial participation
* Medical contraindications for general anesthesia, craniotomy, or surgery.
* Diagnosis of acute myocardial infarction or cardiac arrest within previous 6 months.
* Dementia
* Other implantable devices such as heart/brain pacemakers
* Participants who rely on ventilators
* Co-morbid conditions that would interfere with study activities or response to treatment, which may include:

  * Life expectancy < 3 years
  * Severe chronic pulmonary disease
  * Seizure within three months prior to enrollment
  * History of uncontrolled seizures
  * Local, systemic acute or chronic infectious illness
  * Life threatening cardiac arrhythmias
  * Severe collagen vascular disorder
* Kidney failure or other major organ system failures History of a neurological ablation procedure.
* Labeled contraindication for MRI.
* History of HIV infection or ongoing chronic infection (such as tuberculosis).
* Pregnant or of child-bearing potential and are not taking acceptable methods of contraception.
* Participation in another investigational device or medication trial
* Excessive pain in the paretic upper extremity (> 5 on a 10-point visual analog scale)
* Excessive spasticity at the paretic elbow, wrist, or digits as defined as a score of > 2 on the Modified Ashworth Spasticity Scale
* Participating in any experimental rehabilitation or drug studies
* Moderate to severe apraxia (< 2.5 on the Alexander scale)
* Received phenol injections to any portion of the paretic upper extremity within the past 12 months
* Other conditions or circumstances that, in the opinion of the investigators, would preclude safe and/or effective participation, including severe skin conditions, and/or other sequelae that may be contraindicated for arm orthosis use as well as personal circumstance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Fugl-Meyer Motor Impairment Score at 4 months | 4 months
  The Fugl-Meyer assessment (FMA) is a stroke specific index for estimating the performance of motor function. Total scores of FMA-Upper limb range from 0-66.
  From: Fugl-Meyer et al. The post-stroke hemiplegic patient: a method for evaluation of physical performance. Scand. J. Rehabil. Med., 1975.
Change from Baseline Action Research Arm Test (ARAT) score at 4 months | 4 months
  The Action Research Arm Test (ARAT) measures specific changes in the arm function in people who sustained cerebral damage resulting in arm weakness. The ARAT consists of 19 items grouped into four subscales: grasp, grip, pinch and gross movements. Each sub scale has items ordered according to ascending difficulty: 0- can not perform any part of the test, 1- performs the test partially, 2- completes the test, but takes abnormally long time, 3- performs the test normally. The sum of all subscales are added to compute the total score. The total score ranges between 0 to 57. The higher score is considered to be better outcome.
  From: Yozbatiran et al. A standardized approach to performing the action research arm test. Neurorehabil. Neural Repair, 2008.
Change from Baseline Motricity Index score at 4 months | 4 months
  The Motricity Index measures strength in the arms and legs after stroke. The weighted score is based on the ordinal 6 point scale of Medical Research Council to measure maximal isometric muscle strength.
  From: Collin and Wade. Assessing motor impairment after stroke: A pilot reliability study. J. Neurol. Neurosurg. Psychiatry, 1990.
Change from Baseline ADL, Hand and Recovery Scales within Stroke Impact Scale, at 4 months | 4 months
  The Stroke Impact Scales assess how having a stroke impacts a person's life. The scale has 8 subscales which ask questions regarding a person's physical limitations, memory and thinking, emotions and mood, ability to communicate, daily activities, mobility at home and in the community, use of hand most affected by stroke, and ability to participate in meaningful life activities. Each subscale item is rated on a scale from 5-1 (5= None of the time, 4=a little of the time, 3=Some of the time, 2=Most of the time, 1=All of the time). ADL = activities of daily living.
  From: Duncan et al. The Stroke Impact Scale Version 2.0 : Evaluation of Reliability, Validity, and Sensitivity to Change. Stroke, 1999.

SECONDARY OUTCOMES:
Change from Baseline Braden skin health score at 4 months | 4 months
  The Braden scale predicts pressure sore risk. The Braden score consists of 6 categories: sensory perception, moisture, activity, mobility, nutrition and friction. The score ranges from 6-23 with lower scores indicating a higher risk.
  From: Bergstrom et al. The Braden Scale for Predicting Pressure Sore Risk. Nurs. Res. 36(4): 205-210. 1987.

CONTACTS AND LOCATIONS:
Overall Officials: Mijail Serruya, MD, PhD, Principal Investigator — Dr.
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data are available. The individual participant data comprises those that underlie the results reported in the first article describing outcome measures after deidentification. Other documents available are the Study Protocol and the Analytic Code.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The data will be available beginning 3 months and ending 5 years following publication of the first manuscript summarizing outcome measure results.
Access Criteria: The data is available to researchers who provide a methodologically sound proposal to achieve the aims of the approved proposal. Proposals should be directed to Mijail.Serruya@jefferson.edu . To gain access, data requestors will need to sign a data access agreement. Data will be available for 5 years at a third-party website:
URL: https://doi.org/10.5281/zenodo.5885015